CLINICAL TRIAL: NCT03957109
Title: Influence of Anesthesia Methods on Surgical Outcomes and Renal Function in Retrograde Intrarenal Stone Surgery: a Prospective, Randomized Controlled Study
Brief Title: Influence of Anesthesia Methods on Surgical Outcomes and Renal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-2015-75
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2019-05

CONDITIONS: Kidney Calculi
MeSH Terms: conditions — Kidney Calculi | interventions — Anesthesia, General; Anesthesia, Spinal

ARMS (2):
- general anesthesia (Other): general anesthesia
  Interventions: Procedure: general anesthesia
- spinal anesthesia (Other): spinal anesthesia
  Interventions: Procedure: general anesthesia

INTERVENTIONS:
Procedure: general anesthesia
  Other Names: spinal anesthesia

SUMMARY:
Patients who underwent retrograde intrarenal surgery (RIRS) were randomly allocated to general anesthesia (GA) or spinal anesthesia (SA) groups. Renal function was assessed using estimated glomerular filtration rate, and relative renal function was evaluated using nuclear medicine tests. Maneuverability and accessibility were evaluated after every surgery. We analyzed the influence of anesthesia methods on surgical outcomes and renal function in retrograde intrarenal surgery in a prospective, randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* older than 20 years with renal stones greater than 10 mm

Exclusion Criteria:

* patients who have urologic anatomical abnormalities
* patients with ASA status ≥ grade III, a contraindication for spinal anesthesia or RIRS, or unexpected intraoperative renal injury

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-02-10 (Actual)

PRIMARY OUTCOMES:
Renal function change according to anesthesia method | prior to procedure, and at 3 months after the procedure.
  using nuclear medicine tests with diethylenetriamine pentaacetic acid (99m Tc-DTPA)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kwon O, Lee JM, Park J, Cho MC, Son H, Jeong H, Ryang SH, Cho SY. Influence of anesthesia methods on surgical outcomes and renal function in retrograde intrarenal stone surgery: a prospective, randomized controlled study. BMC Anesthesiol. 2019 Dec 23;19(1):239. doi: 10.1186/s12871-019-0901-9. PMID 31870417